CLINICAL TRIAL: NCT07315763
Title: Polyvagal Informed Group Skills Training for Body Awareness and Managing Emotions for People Living With Obesity
Brief Title: Group Skills Training for Body Awareness and Managing Emotions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Holloway University (Other)
Collaborators: Ashford and St. Peter's Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Jodie Ferris, Trainee Clinical Psychologist, Royal Holloway University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRAS 356169
Record Dates: First submitted 2025-11-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-10

CONDITIONS: Body Awareness; Obesity; Emotional Regulation
Keywords: Body awareness; Specialist Weight Management Service; Polyvagal Theory; Emotional regulation; Polyvagal theory in therapy; Single case experimental design; Skills training; Obesity
MeSH Terms: conditions — Obesity; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: All participants receive the same intervention/treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline Phase (No Intervention): Participants will be randomized to a 2 or 3 week baseline phase.
- Intervention Phase (Experimental): The skills training intervention phase will begin immediately following the individual's baseline phase. The intervention is a group polyvagal theory-informed skills training. The skills training phase is six sessions of polyvagal theory-informed skills training delivered in a group that will take place over nine weeks (three weekly sessions and three fortnightly). Each session will be two hours long. The group will focus on understanding the autonomic nervous system, respecting changes in physiology as a result of the autonomic nervous system, and learning strategies to enhance body awareness and manage emotions, such as breathing exercises. Participants will be asked to practice techniques in sessions and applied independently between sessions with the chance to feedback on the application of ideas and techniques each session.
  Interventions: Behavioral: Polyvagal informed skills training group
- Follow-up Phase (No Intervention): After participants have completed the group skills training, there is a 4 week follow-up phase. During this phase, there is no intervention but participants will continue practicing learned techniques independently.

INTERVENTIONS:
Behavioral: Polyvagal informed skills training group — Research has found a connection between obesity and challenges in managing emotions, including emotional eating (Fernandes et al., 2018; Willem et al., 2019; Konttinen et al., 2019). There is currently a lack of treatments designed to address these issues whilst also promoting a curious and accepting relationship with the body. This may be particularly important for this group who may have a history of dieting or experience internalised stigma which can create a disconnect between the person and their body, a factor that many existing approaches fail to address, even though it is known to negatively impact health (Puhl et al., 2020). This study aligns with recent shifts in health policy, which move away from focusing solely on weight loss and instead prioritise non-weight-related health outcomes (Hunger et al., 2020). This group skills training, based on Polyvagal Theory (Porges, 1995), is designed to meet these needs.
  Other Names: Group PVTT
  Arms: Intervention Phase

SUMMARY:
The goal of this study is to evaluate the effectiveness of a skills training group informed by polyvagal theory, when delivered in an NHS setting, for those living with obesity. Polyvagal Theory in Therapy encourages individuals to be curious, respect how their nervous system works, and notice and respond to bodily sensations. Research shows that interoception, which is the ability to sense and understand what is happening inside the body such as recognising hunger, pain, or emotions, may be challenging for people in larger bodies. These challenges have been connected to difficulties in managing emotions which may lead to behaviours such as emotional eating. This points to the need for a therapeutic approach that helps people both notice what's happening in their bodies and trust those signals enough to be able to respond in healthy ways. This project will test whether a novel polyvagal informed skills training group can improve body awareness (interoception) and emotional regulation for people within an NHS specialist weight management service using a single case experimental design. Participants will be randomly assigned a baseline period of either 14 or 21 (phase A of the design) using computer-generated randomisation. During this phase, participants will complete outcome measures. The skills training intervention phase (phase B) will begin immediately following the individual's baseline period. The intervention is the six session group polyvagal theory-informed skills training. A four-week follow-up period will follow the skills training group, during which participants will continue to complete the same outcome measures they had used in the first two phases. This phase will help assess whether immediate treatment gains are maintained and/or whether delayed treatment gains occur. Trend analysis within this phase will show whether improvement or decline occurs post-skills training.

DETAILED DESCRIPTION:
This study will be a quantitative multiple baseline study using a within-subjects' single case experimental design. The study will take place over three phases; the baseline phase, the skills training intervention phase and the follow-up phase. For the baseline phase, participants will be randomly allocated a baseline period of either 14 or 21 days using an online random number generator, and the intervention (group skills training) will start immediately after the baseline period ends. The skills training phase is six sessions of polyvagal theory-informed skills training delivered in a group that will take place over nine weeks (three weekly sessions and three fortnightly). The intervention effect will be measured through three daily visual analogue scales and two weekly standardised measures. Outcomes will be compared at the same stages across participants. A four-week follow-up period will take place after the skills training. Participants will complete outcome measures throughout all phases. Participants will be asked to commit to a study lasting up to 16 weeks. The study will take place virtually, where questionnaires will be completed online and the group skills training will take place on an online video platform.

The participants will be patients from Ashford and St Peter's NHS Specialist Weight Management Service. They will be identified and approached by the clinical team during routine clinical contact and if the patient is interested in taking part, consent to share their details with the research team will be gained. Participants will be informed on the nature of the skills training group and provided with a video and information sheet explaining what the group will involve so they are able to decide if they wish to take part.

Participants will complete the University of Rhode Island Change Assessment (URICA) to identify their stage of change (Pre-contemplation, Contemplation, Action or Maintenance) before taking part and those in the pre-contemplation stage will not be included. Participants will be informed of this beforehand and it will be explained that this is to ensure that only those who will be best able to engage and make use of the group skills training attend the group and take part in the study, given the high level of commitment. Participants will also complete a demographics questionnaire asking them to self-report their gender, age category, ethnicity and state any comorbidities including physical health conditions, mental health conditions and neurodiversity. This information will not be used to identify the participants but will be used when considering collective group of participants and the generalisability of the findings.

In all phases, participants will complete a brief daily questionnaire in the form of a four question visual analog scale, asking participants to record the frequency they are noticing and responding to shifts in their body and engaging in an unwanted chosen behaviour, such as emotional eating. The fourth question will only be completed during the intervention and follow-up phase and asks participants to record the frequency of skills practice. Participants will also be asked to complete two short online questionnaires weekly that take up to 15 minutes to complete, the Difficulties in Emotion Regulation Scale and the Multidimensional Assessment of Interoceptive Awareness Version 2.

Participants will take part in a six-session group skills training with a Trainee Clinical Psychologist and qualified Clinical Psychologist under the supervision of the the research supervisor, a Clinical Psychologist and the treatment manual creator via video call, scheduled weekly for the first three sessions and fortnightly for the following three sessions, taking place over a nine-week period. Each session will be two hours long. The group will focus on understanding the autonomic nervous system, respecting changes in physiology as a result of the autonomic nervous system, and learning strategies to enhance body awareness and manage emotions, such as breathing exercises. The content of the sessions will include: introduction to polyvagal theory; application of polyvagal theory to client's difficulties; mapping on the polyvagal ladder; exercises to regulate up the ladder; practicing exercises and mapping on the ladder and summarising and skills training blueprint. Participants will be asked to practice techniques in sessions and applied independently between sessions with the chance to feedback on the application of ideas and techniques each session. Participants will be contacted via mobile phone or email to remind them of the group appointment and to complete daily and weekly questionnaires.

After participants have completed the group skills training, during the four-week follow-up phase, participants will complete a feedback form that will be used to assess the acceptability of the group. During this phase, participants will continue practicing learned techniques and continue to complete the daily and weekly questionnaires. At the end of the study, participants will be provided with a full debrief and signposted to further support if needed.

ELIGIBILITY:
Inclusion Criteria:

* Able to commit to the duration of the study from baseline to end of follow up period (up to 16 weeks)
* Current service user of Specialist Weight Management Programme
* Aged 18-65.
* Good level of English spoken, reading and writing.
* Identified by the University of Rhode Island Change Assessment (URICA) to be in the Contemplation, Action or Maintenance stage of change.
* Access to device with internet connection to complete online questionnaires and with camera for online group sessions.

Exclusion Criteria:

* Identified by the University of Rhode Island Change Assessment (URICA) to be in Pre-contemplation stage of change
* Currently in psychological skills training treatment during the 16-week study period
* History of organic brain injury or cognitive impairment
* Clients presenting with suicidal intent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-27 (Estimated); Primary Completion 2026-01-27 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Body awareness and emotional regulation visual analogue scales (VAS) | 16 weeks maximum, from day 1 of the 2- or 3-week baseline, throughout the 9-week intervention and until last day of the 4-week follow up phase.
  To be completed once per day. Includes three questions asking participants about their body awareness, taking care of body shifts and the frequency of a chosen behaviour. The questions are 'Over the last 24 hours, how many times were you able to recognise shifts in your body?' , 'Over the last 24 hours, how many times did you take care of the shifts in your body? ' and 'Over the last 24 hours, how many times have you engaged in your chosen behaviour?' to rate on a scale of 0-20.

SECONDARY OUTCOMES:
Skills practice visual analogue scale (VAS) | 13 weeks maximum, from day 1 of the 9-week intervention and until the last day of the 4-week follow up phase.
  To be completed once per day. Includes one questions asking participants about frequency of skills practice. The question is 'Over the the last 24 hours, how many times have you practiced the skills you have learnt in the group?' to rate on a scale of 0-20.
Difficulties in Emotion Regulation Scale (DERS) | 16 weeks maximum, from day 1 of the 2- or 3-week baseline, throughout the 9-week intervention and until last day of the 4-week follow up phase.
  To be completed weekly. It is a 36-item a measure designed to assess difficulties in emotion regulation, providing insights into an individual's ability to understand, accept, and manage emotions effectively.
Multidimensional Assessment of Interoceptive Awareness Version 2 (MAIA-2) | 16 weeks maximum, from day 1 of the 2- or 3-week baseline, throughout the 9-week intervention and until last day of the 4-week follow up phase.
  To be completed weekly. The Multidimensional Assessment of Interoceptive Awareness Version 2 (MAIA-2) is a self-report questionnaire. It has 37 items and assesses eight different dimensions of interoceptive awareness.

OTHER OUTCOMES:
The University of Rhode Island Change Assessment (URICA) | To be completed once before starting the day 1 of baseline phase.
  To be completed once before starting the baseline phase. The University of Rhode Island Change Assessment (URICA) is a questionnaire used to assess an individual's readiness to change a problem behaviour and categorises individuals into one of four stages of change: Precontemplation, Contemplation, Action, and Maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Jodie F Ferris, Principal Investigator — Royal Holloway University; Jodie S Vasiliou, C.Psychol., Study Chair — Royal Holloway University; Katie S Ashcroft, DClinPsy, Study Director — Royal Holloway University
Locations (1):
- Ashford and St Peter's Hospital NHS Foundation Trust, Ashford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehling WE, Acree M, Stewart A, Silas J, Jones A. The Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-2). PLoS One. 2018 Dec 4;13(12):e0208034. doi: 10.1371/journal.pone.0208034. eCollection 2018. PMID 30513087
- [Background] Porges SW. Orienting in a defensive world: mammalian modifications of our evolutionary heritage. A Polyvagal Theory. Psychophysiology. 1995 Jul;32(4):301-18. doi: 10.1111/j.1469-8986.1995.tb01213.x. PMID 7652107
- [Background] Puhl RM, Himmelstein MS, Pearl RL. Weight stigma as a psychosocial contributor to obesity. Am Psychol. 2020 Feb-Mar;75(2):274-289. doi: 10.1037/amp0000538. PMID 32053000
- [Background] Konttinen H, van Strien T, Mannisto S, Jousilahti P, Haukkala A. Depression, emotional eating and long-term weight changes: a population-based prospective study. Int J Behav Nutr Phys Act. 2019 Mar 20;16(1):28. doi: 10.1186/s12966-019-0791-8. PMID 30894189
- [Background] Fernandes J, Ferreira-Santos F, Miller K, Torres S. Emotional processing in obesity: a systematic review and exploratory meta-analysis. Obes Rev. 2018 Jan;19(1):111-120. doi: 10.1111/obr.12607. Epub 2017 Oct 10. PMID 29024361
- [Background] Willem C, Nandrino JL, Doba K, Roussel M, Triquet C, Verkindt H, Pattou F, Gandolphe MC. Interoceptive reliance as a major determinant of emotional eating in adult obesity. J Health Psychol. 2021 Oct;26(12):2118-2130. doi: 10.1177/1359105320903093. Epub 2020 Jan 31. PMID 32003234
- [Background] Vasileiou V, Abbott S. Emotional eating among adults with healthy weight, overweight and obesity: a systematic review and meta-analysis. J Hum Nutr Diet. 2023 Oct;36(5):1922-1930. doi: 10.1111/jhn.13176. Epub 2023 Apr 19. PMID 37012653
- [Background] Willem C, Gandolphe MC, Roussel M, Verkindt H, Pattou F, Nandrino JL. Difficulties in emotion regulation and deficits in interoceptive awareness in moderate and severe obesity. Eat Weight Disord. 2019 Aug;24(4):633-644. doi: 10.1007/s40519-019-00738-0. Epub 2019 Jun 26. PMID 31243741

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-10-29): https://cdn.clinicaltrials.gov/large-docs/63/NCT07315763/Prot_SAP_000.pdf
  • Informed Consent Form (2025-10-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT07315763/ICF_001.pdf